CLINICAL TRIAL: NCT04223999
Title: Enhancing Tumor Treating Fields for Recurrent Glioblastoma With Targeted and Individualised Skullremodeling Surgery: A Multi-center Randomized Phase 2 Trial
Brief Title: Improving Tumor Treating Fields Treatment for Brain Cancer Patients With Skullremodeling Surgery (Neurosurgery)
Acronym: OptimalTTF-2
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Anders Rosendal Korshøj (Other)
Collaborators: NovoCure GmbH (Industry); Odense University Hospital (Other); Aalborg University Hospital (Other); Rigshospitalet, Denmark (Other)
Responsible Party: Sponsor-Investigator, Anders Rosendal Korshøj, Principal Investigator, Associate Professor, Aarhus University Hospital
Organization: University of Aarhus (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 150919V1; 68928/1-10-72-214-19 (Other: The Danish Central Region Committee on Health Research Ethics); 658876/1-16-02-277-19 (Other: The Danish Data Protection Agency); 2019081231 (Other: The Danish Medical Agency)
Record Dates: First submitted 2019-11-07; First posted 2020-01-13 (Actual); Last update posted 2023-06-06 (Actual); Status verified 2023-06

CONDITIONS: Recurrent Glioblastoma
Keywords: Recurrent glioblastoma; Glioblastoma; Glioblastom; TTFields; Clinical trial; Phase 2; Skullremodeling surgery; Enhancing tumor treating fields; Optimizing tumor treating fields; tumor treating fields; Skull remodeling surgery; SR-surgery; Brain cancer; Experimental neurosurgery
MeSH Terms: conditions — Glioblastoma; Brain Neoplasms

STUDY DESIGN:
Intervention Model Description: Patients will be randomized 1:1 to one of two study arms to receive either, 1) skullremodeling-surgery, TTFields and best practice medical oncological therapy (interventional arm), or 2) TTFields and best practice medical oncological therapy alone (control arm).
Who Masked: Outcomes Assessor
Masking Description: Skullremodeling surgery prevents the participant, careprovider and investigator to be blinded to the randomization.
  The outcome assessors (statisticians) will be blinded when analysing the data.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): In this arm, trial participants receive the intervention that is being tested, skullremodeling surgery. This is in combination with tumor treating fields and best practice medical treatment.
  Interventions: Procedure: Skullremodeling surgery
- Control (Active Comparator): In this arm, the trial participant receives tumor treating fields and best practice medical treatment.
  This serves as an active comparative control arm to the intervention.
  Interventions: Other: Control

INTERVENTIONS:
Procedure: Skullremodeling surgery — Strategically placed cranial burrholes in order to improve the TTField "dose" focally in the tumor.
  Other Names: SR-surgery
  Arms: Intervention
Other: Control — Tumor treating fields combined with best medical treatment.
  Arms: Control

SUMMARY:
The aim of this trial is to test a new potential treatment, skullremodeling surgery (SR-surgery) combined with tumor treating fields (TTFields), for patients with first recurrence of malignant brain tumor (first recurrence of glioblastoma). Glioblastoma is one of the most malignant cancers.

TTFields is a new treatment for brain cancer (glioblastoma), which is used in additional to surgery (removal of the tumor), chemotherapy and radiation. TTFields work by sending alternating current to the tumor. The current disrupts cell division and thus prevents cancer growths. Electrodes are placed on the scalp and the current is delivered via a small portable battery (1kg). Treatment duration is 18 hours during the day, where the patient can do normal daily activities. The average life expectancy of a newly diagnosed brain cancer patient (glioblastoma) is increased from 15 months to 21 months by adding TTFields.

SR-surgery is a minor and safe procedure, that involves creating small burrholes in the skull over the tumor location. The burrholes are approximately 15 mm in diameter. The burrholes increase the electric current in the tumor by funneling the electricity trough the path of least resistance, since bone hinders the electricity.

The theory is that combining TTFields with SR-surgery we can increase the effect of TTFields and in return increase overall survival for brain cancer patients.

The investigators have recently finished a phase 1 clinical trial, with 15 trial participants, testing the safety and efficacy of our combined treatment. The investigators concluded that TTFields and SR-surgery combined is safe and showed promising results by increasing overall survival with the trial participants.

Therefor we wish to proceed with a phase 2 trial.

Method The investigators aim to include 70 patients with first recurrence of glioblastoma (brain cancer). Each patient will be randomized to one of two treatment arms. Both treatment arms will receive the best current brain tumor treatment. In addition, one arm receives TTF and the other arm TTFields and SR-surgery.

All patients are expected to receive better treatment than current best practice, since TTFields is not standard treatment in Denmark.

The primary aim of the trial is to assess the 12-month overall survival in both groups. The theory is that more trial participants will be alive after 12 months in the group that receives both TTF and SR-surgery.

The trial duration is 36 months with an average expected follow-up of 18 months.

DETAILED DESCRIPTION:
Introduction Tumor treating fields (TTFields) are low-intensity (1-3 v/m) intermediate frequency (200 khz for GBM) alternating fields that disrupt cell division. The treatment is increasingly used as a supplementary modality for patients with glioblastoma (GBM). Recent randomized clinical studies have demonstrated tolerability of TTFields (Optune®, Novocure®) for both newly diagnosed and recurrent GBM and a significant and sustained survival benefit in the former population. Specifically, the addition of TTFields to maintenance temozolomide (TMZ) therapy for newly diagnosed GBM patients, who had completed initial concurrent radio-chemotherapy, resulted in significantly prolonged median progression-free survival (PFS = 6.7 vs. 4.0 months, p<0.001) and median overall survival (OS = 20.9 vs. 16.0 months, p<0.001) compared to maintenance TMZ therapy alone (ef-14 trial) (4). Consequently, TTFields were recently approved by the US FDA and included as a category 1 recommendation in the most recent guidelines from the National Comprehensive Cancer Network (NCCN) for the treatment of newly diagnosed GBM. For recurrent GBM, TTFields monotherapy has been shown to have equivalent efficacy and a superior toxicity profile compared to best practice medical oncological therapy. This led to US FDA approval for this indication in 2011. In addition, a post-hoc analysis of the EF-14 dataset has indicated that the addition of TTFields to 2nd line medical oncological treatment at first disease recurrence leads to an overall survival benefit. Finally, the pride dataset showed that the addition of TTFields to current practice of medical oncological treatment was beneficial.

Recently, the investigators proposed a novel approach to calculate the electrical field distribution induced by TTFields therapy of GBM. The approach utilizes finite element analysis and incorporates personalized MRI data to provide a realistic and individualized estimate of the field intensity distribution, which is associated with the antimitotic efficacy of the treatment. Using this approach, the investigators showed that targeted skull-remodeling surgery, e.g. craniectomy or multiple burr-holes, can provide a substantial and highly focused enhancement (~100%) of the median field intensity in supratentorial tumors, while leaving the field distribution in healthy tissues unaffected.

These results support the theoretical rationale that small and clinically feasible craniectomies may improve the clinical efficacy of TTFields for cerebral hemispheric tumors without compromising patient safety. Based on these findings, the investigators recently concluded an open-label, single arm, prospective phase 1 trial (NCT02893137) to investigate safety and feasibility of SR-surgery with TTFields and best practice neuro-oncological therapy for recurrent GBM. The trial was active from December 2016 to May 2019. The planned total number of patients was fifteen. Eligibility criteria included age > 18 years, first recurrence focal supratentorial GBM (RANO), and KPS ≥ 70. Patients were right-censored for OS and PFS at the time of analysis and excluded upon progression, death, SUSARs, or unacceptable AEs. The primary endpoint was toxicity (CTCAEv4.0). The secondary endpoints were OS, PFS, PFS rate at six months (PFS6), objective response rate (ORR) based on the iRANO criteria (14), quality of life (QoL), Karnofsky performance score (KPS), and steroid dose.20 patients were screened, 2 declined, and 3 had KPS < 70. Of the 15 enrolled patients, 4 were excluded prior to TTFields due to radionecrosis/non-recurrence, post-op infection, neurodeficit and withdrawal of consent, respectively. All included patients (11 male and 2 female) had GBM IDH-wt tumors (4 MGMT-methylated). Median KPS was 90 (range 70-100) and median age 57 years (range 39 to 67). All patients received maximum safe resection at recurrence (4 had no residual tumor (RANO), 5 non-measurable disease, and 2 measurable disease). 9 patients received adjuvant bevacizumab monotherapy and 2 temozolomide rechallenge. The mean skull-defect area was 10.6 cm2 (range 7 to 37 cm2) and the median field enhancement 43 % (range 25 to 59%). The median follow-up duration was 10 months and the median TTFields compliance 90% (range 48 to 98%). We observed no SUSARs, no grade 4/5 SAEs, 12 grade 3 SAEs (6 generalized seizures in patients with known epilepsy, 1 post-op infection, 1 diarrhea, 1TIA, 1 fatigue, 1 headache and 1 DVT). The most common grade AE 1-2 was headache 60% CI95%= [32; 84], fatigue 53%, CI95%= [27; 79], skin rash 47%, CI95%= [21; 73], and nausea 40%, CI95%= [16; 68].

Regarding survival results were PFS6 was 64%, CI95%= [35; 85], PFS= 8.8 months, CI95%= [6.2; 13.2], OS= 15.0 months, CI95%= [9.6;16.2], and OS12= 64%, CI95%= [35;85]. One patient had complete response during TTFields. Based on these results, the investigators concluded that skull-remodelling surgery incl. craniectomy is not associated with additional toxicity in combination with TTFields and best practice medical oncological treatment and holds promising potential for improving TTFields outcome by focally enhancing the field intensity in the tumor. The proposed phase 2 trial aims to validate this hypothesis in a randomized comparative setting.

METHODS AND ANALYSIS Trial design The study is designed as an investigator-initiated, prospective, multi-center, multi-national, randomized, minimax two-stage, comparative, phase 2 trial, investigating superior efficacy of the intervention. Patients randomized to the control arm will receive TTFields plus best physician's choice medical oncological treatment (BPC treatment) and patients in the interventional arm will receive SR-surgery in addition to TTFields and BPC treatment. The trial will enroll an expected sample size of 70 patients from 4-6 scandinavian countries with Aarhus University Hospital, Denmark, as the Sponsor and coordinating site. The primary outcome will be overall survival at 12 months (OS12) and the trial is designed to detect a 20% increase in OS12 in the interventional arm compared to control (from 40% in the control arm to 60% in the interventional arm). Secondary outcomes will include progression-free survival (PFS), quality of life (QoL), clinical performance, and objective response rate (ORR). Interim futility analysis will be conducted after 12 months follow-up of the first 52 patients. The trial will be stopped at interim analysis if the OS12 months is lower in the control arm compared to the interventional arm. The trial design and data reporting is in accordance with the consort 2010 statement, the gnosis standards for neuro-oncology trials, recent RANO recommendations for phase 2 trial design in neuro-oncology, and general recommendations for phase 2/3 trial design (16-19). The study will be performed in the period march 2020 to march 2023. The inclusion period is expected to be the first 24 months of the trial.

Participants Seventy (70) patients with progressive GBM according to RANO criteria will be enrolled. Potential trial participants will be identified at an institutional multidisciplinary neuro-oncological tumor boards and subsequently referred for eligibility screening. All inclusion scans are assessed by a trained neuroradiologist. Patients who are immediately ineligible, e.g. due to poor performance status, multifocal disease, significant comorbidity, evidence of extracranial primary tumor, or other excluding circumstances, will not be referred for screening.

Experimental intervention Patients will be randomised 1:1 to one of two study arms to receive either, 1) SR-surgery, TTFields and best practice medical oncological therapy (interventional arm), or 2) TTFields and best practice medical oncological therapy alone (control arm). Best practice treatment will typically also include maximum safe resection. Since the intervention (SR-surgery) is only effective during TTFields therapy, TTFields will continue until 1) patient exclusion from the trial, 2) occurrence of a suspected unexpected serious adverse reaction (SUSAR) related to the intervention, or 3) ethical or medical safety contraindication for further TTFields therapy determined by the investigators. This means that treatment may continue beyond progression, as long as active treatment is indicated, and in some cases as compassionate use.

Sample size and statistical considerations The sample size calculations were based on a randomized, comparative, minimax two-stage design and the binomial primary outcome of OS12 for the patient population treated per protocol, i.e. for whom TTFields therapy was initiated. This means that patients excluded prior to TTFields therapy initiation are not included in the primary outcome analysis. Therefore, additional patients may be enrolled to ensure that the planned sample receives active TTFields treatment. The aim of the trial is to determine whether the intervention is superior to control and thus worthy of further phase 3 investigation. The expected OS12 in the control arm is set to 40% based on the EORTC 26101 trial, in which patients with first recurrence of GBM were treated with lomustine monotherapy or lomustine/bevacizumab combination therapy. The trial showed an OS12 of approximately 30% and we therefore set the expected level of OS12 to be slightly above this threshold given the fact that TTFields is added to the treatment which otherwise represents recommended practice. There are no current studies providing accurate OS12 estimates for a population comparable to the study control arm and we therefore based the estimate on an expected benefit of 10% from TTFields alone compared to EORTC 26101. Setting the probabilities of false-positive and false-negative trial results to α = 0.15 and 1-β = 0.80, respectively, and defining the expected target level of OS12 to be OS12 = 0.6, i.e. a 20% absolute increase (and 50% relative increase) compared to the control arm, we calculated a maximum sample size of n = 42 patients in each arm (total n = 84) and an expected total sample size (en = 69.8). The expected sample size en is calculated as en = n1 × pet0 + n × (1 - pet0), where n1 = 52 is the collective sample size of both groups at interim (stage 1) analysis, pet0 = 0.44 is the probability of early futility termination. The numbers are based on the given statistical parameters and a two-stage minimax design as given in sh jung 2018. Interim futility analysis will be conducted after endpoint assessment of 52 patients and the trial will be terminated if the experimental arm performs worse than the control arm. In this case the futility criterion will be defined as OS12experimental < OS12control and this conclusion will determine futility at marginal power and significance levels of 1-β* = 0.80 and of α* = 0.20, respectively. If the trial is not terminated at interim stage 1 analysis, the trial will proceed to enroll a total of 84 patients and terminate when the final OS12 endpoint data have been obtained for all patients.

The secondary outcome measures of hazard rate ratios of PFS and OS will be tested using the log-rank test at the 0.05 alpha level. Time-to-event endpoints will be estimated from the time of randomization. Toxicity and adverse events will be reported using absolute numbers and appropriate risk estimates. Final analysis will be conducted when all patients have been excluded or censored, e.g. due to end-of-trial, or loss-to-follow-up. Subgroup analysis based on prognostic factors will be performed, incl. analysis of patient characteristics in each arm and identification of characteristics of potential responders to the intervention. This will also include a correlation analysis between the calculated field distribution and outcome estimates. Analyses will be based on both the intent-to-treat population and the population proceeding to active therapy (per protocol), i.e. At least four weeks of active TTFields therapy with ≥75% average compliance.

Randomisation and blinding Patients will be randomised immediately upon enrollment in the trial, i.e. prior to initial surgery. Randomisation will be performed using randomization.com and patients will be randomised in a 1:1 ratio to receive TTFields and best practice medical oncological treatment w/o skull remodeling surgery. The study endpoint assessment committee will be blinded to the intervention. Local principal investigators, co-investigators and sub-investigators will not be blinded, as optimal array planning will require knowledge about skull-remodeling surgery. The operating surgeon performing the skull-remodeling surgery will not be blinded. Patients will not be blinded, as it will be possible for the patient to feel the skull configuration and thereby determine whether SR-surgery was performed.

Risks and safety precautions General safety considerations concerning Optune® therapy are outlined in the related technical and safety material provided by Novocure®. In general, TTFields therapy is regarded a safe and recognized treatment for GBM. The most common adverse effect is local skin rash in the area underlying the transducer arrays. The risk of skin rash will be reduced by slightly moving the arrays during regular array changes. Skin rash may be treated with topical corticosteroids, more frequent electrode replacement and short pauses in TTFields therapy, if needed. The risk of brain injury due to the skull remodeling aspect of surgery is minimal, as the entire operation is performed extra-durally. Minor craniectomies do not pose a significant risk of mechanical brain injury. For larger craniectomies, external protective headgear, such as a cap with mechanical reinforcement over the unprotected brain area, may be used to reduce the risk of traumatic brain injury after craniectomy. In the case of post-operative infection or impaired wound healing, antibiotic therapy will be administered. If needed, surgical revision/debridement of the wound and potentially removal of the bone flap may be performed. In such cases, the patient may proceed to receive or continue TTFields therapy at an appropriate time, if it is in the patient's best interest. TTFields therapy following removal of the infected bone flap may be accepted even if the craniectomy size exceeds 30 cm2. In all cases, the decision whether to continue with TTFields therapy after surgery will be based on careful consideration of the expected safety and benefit for the patient. All participants will be advised of situations and adverse events, in which medical attention is required. Investigators or properly trained medical personnel will be available for immediate attention or medical advice specific to the treatment or protocol. Patients will receive contact information to the device support specialist, whom they may contact in case of technical problems or considerations.

Monitoring and quality control The project will comply with international guidelines good clinical practice (ICH-GCP and ds/en iso 14155:2012. Clinical investigation of medical devices for human subjects - good clinical practice) and be monitored by the local contract research organization (CRO). Source data, verification of consent, and handling of adverse events and near-miss incidents will be subject to 20% sampled monitoring. Full access to all source data, incl. patient records, will be granted in relation to trial inspection by the relevant national competent authorities. Experimental "waivers" from the protocol will be registered in the project trial master file and reported to the relevant authorities. Changes to the protocol will be submitted for approval by the relevant authorities in accordance with GCP guidelines and regulations.

Dissemination All results will be published in peer-reviewed international scientific journals and presented at international scientific conferences, regardless of academic conclusions. Positive, negative, and inconclusive results will be publicly available.

ELIGIBILITY:
Inclusion Criteria:

1. age 18 years or older
2. progressive GBM based on the RANO criteria and whole brain MRI according to the consensus recommendations for a standardized brain tumor imaging protocol in clinical trials , not older than 4 weeks from the assessment
3. estimated survival≥ 3 months
4. supratentorial tumor location
5. focal disease in the vicinity of the previously known tumor or resection cavity,
6. KPS≥70
7. ability to comply with TTFields treatment
8. eligibility for diagnostic or therapeutic neurosurgery and subsequent best practice oncological therapy,
9. tumor characteristics indicating significant expected benefit from feasible craniectomy or SR-surgery combined with TTFields i.e. (a) focal tumor and (b) most superficial border of tumor or resection cavity closer than 2 cm from brain surface
10. use of validated anticonception for fertile female participants in concordance with guidelines provided by the danish health and medicines authority,
11. signed written consent form

Exclusion Criteria:

1. pregnancy or nursing (fertile female participants will be required to take a validated pregnancy test for evaluation of pregnancy)
2. infra-tentorial tumor
3. implanted pacemaker, defibrillator, deep brain stimulator, other implanted electronic devices in the brain, or documented clinically significant arrhythmia
4. uncontrollable symptomatic epilepsy refractory to standard medication
5. contraindications for skullremodeling surgery, e.g.bleeding diathesis or severe infection
6. significant co-morbidities, i.e. (a)significant liver function impairment (alt >210 u/l for men and > 135 u/l for women or total bilirubin >25umol/l), (b)significant renal impairment (serum creatinine > 1.7 mg/dl= 150 umol/l), (c)coagulopathy (inr> 1.8 or aptt > 57s), (d) thrombocytopenia (platelet count < 100 x 103/μl =100 x 109/l), (e) neutropenia (anc< 1.5 x 103/μl =1.5 x 109/l), (f) anemia ( hb < 10 g/l= 6.0 mmol/l)
7. severe cognitive impairment
8. active participation in another therapeutic interventional clinical trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2020-10-01 (Actual); Primary Completion 2024-03-01 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
OS12 | 12 months from the time of randomization.
  12-month overall survival.

SECONDARY OUTCOMES:
Median OS | From date of randomization until the date of death from any cause, assessed up to 60 month.
  Median overall survival.
Median PFS | From date of randomization until the date of first documented progression, assessed up to 36 months.
  Median progression-free survival.
OS24 | 24 months from the time of randomization.
  24-month overall survival
OS36 | 36 months from the time of randomization.
  36-month overall survival
PFS6 | 6 months from the time of randomization
  6-month progression-free survival
ORR | Assessed every 3. month, up to 36 months or death, whichever comes first.
  Overall objective response rate assessed by modified RANO criteria
Standardised and verified quality of life assessment questionnaires (QLQ-C30 and QLQ-BN20) for cancer and brain tumor patients. | Assessed at inclusion and every 3. month, assessed up to 36 months or death, whichever comes first.
  Standardised and verified questions related to quality of life to cancer and brain tumor patients. Quality of life is rated by the patients own thoughts about the current situation and future and also the presence or absence of the most common symptoms in cancer and brain tumors. Rated from a scale 1-4 (none to a lot) and 1-7 scale (very poor to very good).
Steroid dose | From the time of inclusion and every 3. month, assessed up to 36 months or death, whichever comes first.
  Cumulative corticosteroid usage
KPS | From time of inclusion and every 3. month, assessed up to 36 months or death, whichever comes first.
  Assessing KPS.
AE | From time of inclusion and every 3. month, assessed up to 36 months or death, whichever comes first.
  Adverse events / Safety. All adverse events observed by personnel or reported by trial participant.

CONTACTS AND LOCATIONS:
Overall Officials: Anders R Korshøj, MD, PhD, Principal Investigator — Aarhus University Hospital
Locations (1):
- Nikola Mikic, Aarhus, Denmark

IPD SHARING:
Plan to Share IPD: No
All data published will be available upon request. Study protocol will be published.